CLINICAL TRIAL: NCT06002685
Title: Effects of Attachment-Based Intervention on Low-Income Latino Children's Emerging Health Outcomes
Brief Title: Partners in Children's Health (CSN): A Randomized Trial of an Attachment Based Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Johns Hopkins University (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Lisa Berlin, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00103602
Record Dates: First submitted 2023-06-06; First posted 2023-08-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Disease; Inflammation; Insufficient Sleep; Digestive Disease; Skin Conditions; Body Mass Index; Infections; Allergies; Congestion; Antibiotic Use; Overweight and Obesity
MeSH Terms: conditions — Respiration Disorders; Inflammation; Sleep Deprivation; Digestive System Diseases; Skin Diseases; Infections; Hypersensitivity; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A 2-group, pre-and post-test experimental design (N = 260; 130 in each group) will be employed. All eligible mother-child dyads will be randomly assigned to receive the intervention, Attachment Biobehavioral Catch- up (ABC),or the control, Home-Book-of-the- Week (HBOW). Assessments will take place in the participant's home and on the phone.
Who Masked: Outcomes Assessor
Masking Description: 2 tasks will be coded by research assistants masked to assigned intervention condition.
  Child Stress Regulation: Using video-recorded data collected at Times 1 and 2, blinded coders will rate the child's emotion regulation strategies in the context of mild stressors. Coders will use the Laboratory Temperament Assessment Battery (Lab-TAB) to rate the presence/absence of the following behaviors every 5 seconds: looks to mother, communicative gestures, looks to environment; and self-stimulation. In keeping with our own and others' previous data reduction in this domain, we will compute two proportion-score composites for mother-oriented regulation and self-soothing regulation. Coders will rate children's emotional re-activity every 5 seconds to analyze emotional reactivity as a covariate.
  Sensitive Parenting Behaviors: At Times 1 and 2, blinded coders will collect observational assessments of sensitive parenting behaviors in 3 contexts: (a) play, (b) child distress, and (c) feeding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment and Biobehavioral Catch-up (ABC) program (Experimental): The ABC program consists of 10 1 -hour home-based sessions delivered by a trained parent coach. Each session includes the mother and her child together and addresses a specific topic.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-Up
- Home-Based Book-of-the-Week (HBOW) program (Active Comparator): The HBOW program consists of 10 English/Spanish developmentally appropriate books hand-delivered weekly to the mothers. A trained RA will utilize a standard set of questions to ask about the mother's and child's well-being.
  Interventions: Other: Home-Based Book-of-the-Week

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-Up — The ABC program consists of 10 one-hour home-based sessions delivered by a trained parent coach. Each session includes the mother and her child together and addresses a specific topic. Principal intervention activities include a discussion of basic attachment principles, guided practice of new parenting behaviors, and a review of video clips from previous sessions to help reinforce parenting targets. The parent coach promotes (a) nurturance, especially in response to distress; (b) following the child's lead with delight; and (c) avoiding frightening caregiving behavior. As specified by the ABC protocol, any/all other family members will be invited to observe or participate in each ABC session Each full-time ABC parent coach will serve 8 to 10 families at a time (i.e., complete 8-10 hourly ABC visits per week).
  Other Names: ABC
  Arms: Attachment and Biobehavioral Catch-up (ABC) program
Other: Home-Based Book-of-the-Week — The HBOW program is an active control condition developed by PI Berlin. It consists of 10 English/Spanish developmentally appropriate books hand-delivered weekly to the mothers. During each of the 10 weeks, a trained RA will visit each HBOW mother to drop off the book and to ask briefly about the mother's and child's well-being (using a standard set of questions). Thus, this condition will parallel the intervention condition in duration (number of weeks) and structure, although it will be less intensive in terms of participant contact time per visit.
  Other Names: HBOW
  Arms: Home-Based Book-of-the-Week (HBOW) program

SUMMARY:
The goal of this randomized controlled trial is to evaluate the impacts of an attachment-based intervention (Attachment Biobehavioral Catch-Up (ABC) and Home Book-of-the-Week (HBOW) program on emerging health outcomes (i.e., common childhood illnesses, body mass index, and sleep) in low-income Latino children (N=260; 9 months at enrollment). It is hypothesized that children randomized to ABC will have better health outcomes in comparison to the HBOW control group.

DETAILED DESCRIPTION:
The proposed RCT will test the impacts of the Attachment Biobehavioral Catch-up (ABC) intervention program on child health outcomes. A total of 260 male and female infants will be enrolled in this study, with an age range of 8-12 months (infant) and 13 months- 23 months (toddler). This study will enroll primiparous and multiparous mothers who identify as Latina, speak English or Spanish, and have a 9-month-old child enrolled in Medicaid at the start of the study. Participants will be recruited in collaboration with the Children's Medical Practice (CMP) at Johns Hopkins Bayview Medical Center and matriculated on a rolling basis. Each participant will participate for approximately 15 months; the time required to complete the Time 1 assessment, either 10-week condition, and the two post-intervention assessments. The entire study is anticipated to be completed in 5 years. This RCT will test maternal sensitivity and child stress regulation as mediators of intervention effects. It will also examine the extent to which sociocultural factors moderate the effects of ABC. Behavioral methods and procedures will include surveys/questionnaires, audio/video recordings, individual or group behavioral observations, psychosocial or behavioral interventions, and other psychosocial or behavioral procedures. This RCT is powered to detect small-medium intervention effects (Cohen's d's= 0.35 - 0.50). These effect sizes align with previous studies, which have shown small to large effects on maternal sensitivity (d's = 0.23 - 0.77) and small to medium effects on main and moderated child behavioral stress regulation (d's= 0.15 - 0.48) and child physiological (cortisol) regulation, via maternal sensitivity (d=-0.36). For .80 power or higher and a two-tailed significance level of .05, power analyses performed using Optimal Design, Webpower, and Gpower software indicated a post-attrition sample size of N=221 will adequately detect main, mediated, and moderated effects of comparable size. Analyses will be conducted in SAS 9.4, SPSS 25.0, and Mplus 8 and will include regression and structural equation models. Missing data will be accommodated using multiple imputations and/or full information maximum likelihood (FIML) and estimators that are robust to non-normality when missing data are present (e.g., MLR). Data safety monitoring will be conducted by the Principal Investigators and the external Data Safety and Monitoring Board, who will review adverse events, enrollment numbers, procedure reports, raw data, outcomes, preliminary analyses, and other data which will be completed on an ongoing basis and reported to the IRB and a sponsor. Study findings stand to inform the nature and timing of preventive interventions to reduce health disparities that disproportionately impact Latino families and will advance understanding of early social influences that promote health development across the lifespan.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers
* Identify as Latina
* Speak English or Spanish
* Primiparous and multiparous
* Have a 9-month-old child enrolled in Medicaid

Exclusion Criteria:

* Children born prematurely (gestational age < 37 weeks)
* Children who have major complex medical conditions (e.g., heart or autoimmune conditions) that could interfere with participation in intervention sessions and/or research assessments.

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Common Childhood Illnesses (cough, runny nose, prescribed antibiotic use) | This data will be gathered at Time 1 (9 months).
  This outcome will be assessed via maternal report and review of the child's electronic health record (EHR). Using the International Classification of Primary Care, mother's responses will be coded into one of five categories reflecting the frequency of general illnesses, respiratory illnesses, digestive illnesses, skin conditions, and antibiotic use.
Common Childhood Illnesses (cough, runny nose, prescribed antibiotic use) | This data will be gathered at Time 2 (15 months).
  This outcome will be assessed via maternal report and review of the child's electronic health record (EHR). Using the International Classification of Primary Care, mother's responses will be coded into one of five categories reflecting the frequency of general illnesses, respiratory illnesses, digestive illnesses, skin conditions, and antibiotic use.
Common Childhood Illnesses (cough, runny nose, prescribed antibiotic use) | This data will be gathered at Time 3 (24 months).
  This outcome will be assessed via maternal report and review of the child's electronic health record (EHR). Using the International Classification of Primary Care, mother's responses will be coded into one of five categories reflecting the frequency of general illnesses, respiratory illnesses, digestive illnesses, skin conditions, and antibiotic use.
Rapid Weight Gain | This data will be gathered at Time 1 (9 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Rapid Weight Gain | This data will be gathered at Time 2 (15 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Rapid Weight Gain | This data will be gathered at Time 3 (24 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Expressive Speech Delay | This data will be gathered at Time 1 (9 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Expressive Speech Delay | This data will be gathered at Time 2 (15 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Expressive Speech Delay | This data will be gathered at Time 3 (24 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Other Pediatric Health Problem(s) | This data will be gathered at Time 1 (9 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Other Pediatric Health Problem(s) | This data will be gathered at Time 2 (15 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Other Pediatric Health Problem(s) | This data will be gathered at Time 3 (24 months).
  This outcome will be assessed through a review of the children's Electronic Health Record.
Low Grade Inflammation | This data will be gathered at Time 3 (24 months).
  This outcome will be assessed via markers of C-reactive protein (CRP) and interleukin-6 (IL-6) through a collection of blood spots using a traditional finger-prick. Blood spot collection is required at the 24-month pediatric well-child visit for all Baltimore City residents.
Body Mass Index | This data will be gathered at Time 1 (9 months).
  This outcome will be collected by an RA by measuring the child's length and weight. Length will be measured using a measurement board. All weight measurements will be obtained in a clean diaper utilizing an infant scale (Seca 374). In addition to this, the child's EHR will be reviewed to extract length and weight data. BMI scores will be calculated using the World Health Organization sex-specific BMO-for-age growth charts per recent guidance for research on early obesity risk.
Body Mass Index | This data will be gathered at Time 2 (15 months).
  This outcome will be collected by an RA by measuring the child's length and weight. Length will be measured using a measurement board. All weight measurements will be obtained in a clean diaper utilizing an infant scale (Seca 374). In addition to this, the child's EHR will be reviewed to extract length and weight data. BMI scores will be calculated using the World Health Organization sex-specific BMO-for-age growth charts per recent guidance for research on early obesity risk.
Body Mass Index | This data will be gathered at Time 3 (24 months).
  This outcome will be collected through mothers reports about their children's current length and weight. In addition to this, the child's EHR will be reviewed to extract length and weight data. BMI scores will be calculated using the World Health Organization sex-specific BMO-for-age growth charts per recent guidance for research on early obesity risk.
Sleep: Age 9 months | Sleep data will be gathered at Time 1 (age 9 months).
  This outcome will be assessed using actigraphy and maternal report. A MotionWatch-8 actigraph will be placed on the child's ankle for continuous (24-hour) recording of body motility in 1-minute epochs. Values will be aggregated over 5 days to assess day/night sleep start times, minutes awake, and sleep efficiency. A total of 7 days of data will be collected to account for missing days that might occur. After the 7 days, an RA will pick up the watch from the mother. An RA will text the mothers a URL to a brief sleep diary for the collection of subjective reports on sleep variations.
Sleep: At 9 months | Sleep data will be gathered at Time 1 (at 9 months).
  An RA will also administer a 33-item Brief Infant Sleep Questionnaire-Revised (BISQ-R) to assess general sleeping habits including bedtime routines, location(s) when the child sleeps, child mood upon wakening, and respondent (maternal) perception of the extent to which the child's sleep is problematic.
Sleep: Age 15 months | Sleep data will be gathered at Time 2 (age 15 months).
  This outcome will be assessed using actigraphy and maternal report. A MotionWatch-8 actigraph will be placed on the child's ankle for continuous (24-hour) recording of body motility in 1-minute epochs. Values will be aggregated over 5 days to assess day/night sleep start times, minutes awake, and sleep efficiency. A total of 7 days of data will be collected to account for missing days that might occur. After the 7 days, an RA will pick up the watch from the mother. An RA will text the mothers a URL to a brief sleep diary for the collection of subjective reports on sleep variations.
Sleep: At 15 months | Sleep data will be gathered at Time 2 (at 15 months).
  An RA will also administer a 33-item Brief Infant Sleep Questionnaire-Revised (BISQ-R) to assess general sleeping habits including bedtime routines, location(s) when the child sleeps, child mood upon wakening, and respondent (maternal) perception of the extent to which the child's sleep is problematic.
Sleep: Age 24 months | Sleep data will be gathered at Time 3 (age 24 months).
  This outcome will be assessed using actigraphy and maternal report. A MotionWatch-8 actigraph will be placed on the child's ankle for continuous (24-hour) recording of body motility in 1-minute epochs. Values will be aggregated over 5 days to assess day/night sleep start times, minutes awake, and sleep efficiency. A total of 7 days of data will be collected to account for missing days that might occur. After the 7 days, an RA will pick up the watch from the mother. An RA will text the mothers a URL to a brief sleep diary for the collection of subjective reports on sleep variations.
Sleep: At 24 months | Sleep data will be gathered at Time 3 (at 24 months).
  An RA will also administer a 33-item Brief Infant Sleep Questionnaire-Revised (BISQ-R) to assess general sleeping habits including bedtime routines, location(s) when the child sleeps, child mood upon wakening, and respondent (maternal) perception of the extent to which the child's sleep is problematic.

OTHER OUTCOMES:
Maternal Sensitivity during Semi-Structured Play | This data will be collected at Time 1 (9 months).
  This outcome will be assessed with a 15-minute "Three Bag" interaction. The mother will be given vague instructions involving 3 numbered cloth bags, each containing one or more standard, age-graded toys or books, asking that the child spend some time with each. The mother will be informed that she can play or help however she wants. Coders will use the well-established Parent-Child Interaction Rating Scales to assign a global 5-point score for the mother's sensitivity/responsiveness, intrusiveness, and positive regard. This will be video-recorded for subsequent coding by trained, reliable, and blinded coders.
Maternal Sensitivity during Semi-Structured Play | This data will be collected at Time 2 (15 months).
  This outcome will be assessed with a 15-minute "Three Bag" interaction. The mother will be given vague instructions involving 3 numbered cloth bags, each containing one or more standard, age-graded toys or books, asking that the child spend some time with each. The mother will be informed that she can play or help however she wants. Coders will use the well-established Parent-Child Interaction Rating Scales to assign a global 5-point score for the mother's sensitivity/responsiveness, intrusiveness, and positive regard. This will be video-recorded for subsequent coding by trained, reliable, and blinded coders.
Maternal Sensitivity to Child Distress | This data will be collected at Time 1 (9 months).
  This will be assessed in the context of age-graded mild stressors designed to elicit child fear or frustration, all of which have been well-validated. Before each stressor, there will be a 3-minute "baseline" period during which the child will view a neutral video. At Time 1, the stressors will consist of a 4-minute novel toy approach and 3-minute barrier task. At Time 2, the stressors will consist of a 2-minute mask task and a 3-minute barrier task. Following each stressor, there will be a 2-minute child-mother "reunion" when the mother is free to interact with her child however she wants. Mothers will be asked ahead of time not to provide a pacifier or breastfeed during these 2 minutes; after two minutes mothers can interact freely, which will allow researchers to capture mothers' "food to soothe" behaviors. Coders will rate sensitivity to child distress using a 5-point scale. If the child does not display distress, coders will rate the mother's responses to her child's other cues.
Maternal Sensitivity to Child Distress | This data will be collected at Time 2 (15 months).
  This will be assessed in the context of age-graded mild stressors designed to elicit child fear or frustration, all of which have been well-validated. Before each stressor, there will be a 3-minute "baseline" period during which the child will view a neutral video. At Time 1, the stressors will consist of a 4-minute novel toy approach and 3-minute barrier task. At Time 2, the stressors will consist of a 2-minute mask task and a 3-minute barrier task. Following each stressor, there will be a 2-minute child-mother "reunion" when the mother is free to interact with her child however she wants. Mothers will be asked ahead of time not to provide a pacifier or breastfeed during these 2 minutes; after two minutes mothers can interact freely, which will allow researchers to capture mothers' "food to soothe" behaviors. Coders will rate sensitivity to child distress using a 5-point scale. If the child does not display distress, coders will rate the mother's responses to her child's other cues.
Maternal Sensitivity during Feeding | This data will be collected at Time 1 (9 months).
  This outcome will be assessed in terms of maternal responsiveness to child feeding cues and the use of food to soothe child distress, both of which will be observed throughout the home-based assessments. Each home-based assessment will be schedule to include at least one opportunity to observe child feeding./ A set of developmentally and culturally appropriate snack foods will be provided to facilitated standardized observations of mothers' use of food to soothe child distress. Two validated and complementary behavioral coding schemes, the Responsiveness to Child Feeding Cues Scale and the Food to Soothe scheme will be used. This will be video-recorded for subsequent coding by trained, reliable, and blinded coders.
Maternal Sensitivity during Feeding | This data will be collected at Time 2 (15 months).
  This outcome will be assessed in terms of maternal responsiveness to child feeding cues and the use of food to soothe child distress, both of which will be observed throughout the home-based assessments. Each home-based assessment will be schedule to include at least one opportunity to observe child feeding./ A set of developmentally and culturally appropriate snack foods will be provided to facilitated standardized observations of mothers' use of food to soothe child distress. Two validated and complementary behavioral coding schemes, the Responsiveness to Child Feeding Cues Scale and the Food to Soothe scheme will be used. This will be video-recorded for subsequent coding by trained, reliable, and blinded coders.
Child Stress Regulation: Age 9 months | This data will be collected at Time 1 (9 months).
  Video recorded data collected will rate infants' emotion regulation strategies in the context of mild stressors during the above-mentioned three contexts of parenting behaviors. The Laboratory Temperament Assessment Battery will be used to rate the presence/absence of the following 5 behaviors: looks to mother, communicative gestures, looks to the environment, and self-stimulation. A two-proportion score composite will be computed for mother-oriented regulation and self-soothing regulation. Coders will also rate children's emotional reactivity every 5 seconds to analyze emotional reactivity as a covariate. This outcome will be video-recorded for subsequent coding by trained, reliable, and blinded coders.
Child Stress Regulation: Age 15 months | This data will be collected at Time 2 (age 15 months).
  Video recorded data collected will rate infants' emotion regulation strategies in the context of mild stressors during the above-mentioned three contexts of parenting behaviors. The Laboratory Temperament Assessment Battery will be used to rate the presence/absence of the following 5 behaviors: looks to mother, communicative gestures, looks to the environment, and self-stimulation. A two-proportion score composite will be computed for mother-oriented regulation and self-soothing regulation. Coders will also rate children's emotional reactivity every 5 seconds to analyze emotional reactivity as a covariate.
Child Stress Regulation: At 15 months | This data will be collected at Time 2 (at 15 months).
  The child's emotional dysregulation will be assessed by administrating mothers the Infant-Toddler Social and Emotional Assessment (ITSEA). The following three ITSEA subscales will be examined: internalizing, externalizing, and dysregulation. This outcome will be video-recorded for subsequent coding by trained, reliable, and blinded coders.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Berlin, PhD, Principal Investigator — University of Maryland; Natalie Slopen, PhD, Study Chair — Harvard School of Public Health (HSPH); Cathi Propper, PhD, Study Chair — Department of Psychology and Neuroscience at UNC Chapel Hill
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3-5yrs after initial study publications.
Access Criteria: There will be only one master database in which participants' ID numbers and personal identifying information are linked. Only Dr. Berlin and the staff members who are directly involved in the data collection and processing will have access to this database. Electronic data will be stored on a secure network, with password protection such that only authorized users will have access to the file server. Any original data documents such as consent forms will be kept in locked compartments separate from identifying documentation. All electronic and paper files that contain identifying information will be destroyed at the conclusion of the research. Published data will not permit the identification of individuals

REFERENCES:
- [Background] Dozier M, Bernard K. Coaching parents of vulnerable infants: The Attachment and Biobehavioral Catch-Up Approach. Guilford Press; 2019.
- [Background] Berlin LJ, Martoccio TL, Jones Harden B. Improving early head start's impacts on parenting through attachment-based intervention: A randomized controlled trial. Dev Psychol. 2018 Dec;54(12):2316-2327. doi: 10.1037/dev0000592. Epub 2018 Oct 18. PMID 30335427
- [Background] Urquhart A, Clarke P. US racial/ethnic disparities in childhood asthma emergent health care use: National Health Interview Survey, 2013-2015. J Asthma. 2020 May;57(5):510-520. doi: 10.1080/02770903.2019.1590588. Epub 2019 Apr 8. PMID 30958048
- [Background] Kaar JL, Schmiege SJ, Kalkwarf HJ, Woo JG, Daniels SR, Simon SL. Longitudinal Assessment of Sleep Trajectories during Early Childhood and Their Association with Obesity. Child Obes. 2020 Apr;16(3):211-217. doi: 10.1089/chi.2019.0126. Epub 2019 Nov 21. PMID 31750742
- [Background] Berlin LJ, Martoccio TL, Bryce CI, Jones Harden B. Improving infants' stress-induced cortisol regulation through attachment-based intervention: A randomized controlled trial. Psychoneuroendocrinology. 2019 May;103:225-232. doi: 10.1016/j.psyneuen.2019.01.005. Epub 2019 Jan 4. PMID 30716550
- [Background] Cespedes EM, Rifas-Shiman SL, Redline S, Gillman MW, Pena MM, Taveras EM. Longitudinal associations of sleep curtailment with metabolic risk in mid-childhood. Obesity (Silver Spring). 2014 Dec;22(12):2586-92. doi: 10.1002/oby.20894. Epub 2014 Sep 19. PMID 25234485
- [Background] Dowd JB, Zajacova A, Aiello A. Early origins of health disparities: burden of infection, health, and socioeconomic status in U.S. children. Soc Sci Med. 2009 Feb;68(4):699-707. doi: 10.1016/j.socscimed.2008.12.010. Epub 2009 Jan 17. PMID 19152993
- [Background] Meltzer LJ, Pugliese CE. Sleep in young children with asthma and their parents. J Child Health Care. 2017 Sep;21(3):301-311. doi: 10.1177/1367493517712064. Epub 2017 Jun 5. PMID 29119809
- [Background] El-Sheikh M, Buckhalt JA, Granger DA, Erath SA, Acebo C. The association between children's sleep disruption and salivary interleukin-6. J Sleep Res. 2007 Jun;16(2):188-97. doi: 10.1111/j.1365-2869.2007.00593.x. PMID 17542949
- [Background] Hepworth AD, Berlin LJ, Salas K, Pardue-Kim M, Martoccio TL, Jones Harden B. Increasing maternal sensitivity to infant distress through attachment-based intervention: a randomized controlled trial. Attach Hum Dev. 2021 Dec;23(6):953-968. doi: 10.1080/14616734.2020.1834592. Epub 2020 Oct 27. PMID 33108981
- [Background] Worobey J, Lopez MI, Hoffman DJ. Maternal behavior and infant weight gain in the first year. J Nutr Educ Behav. 2009 May-Jun;41(3):169-75. doi: 10.1016/j.jneb.2008.06.005. PMID 19411050
- [Background] Hodges EA, Propper CB, Estrem H, Schultz MB. Feeding During Infancy: Interpersonal Behavior, Physiology, and Obesity Risk. Child Dev Perspect. 2020 Sep;14(3):185-191. doi: 10.1111/cdep.12376. Epub 2020 Jul 14. PMID 34707686
- [Background] Pachter LM, Coll CG. Racism and child health: a review of the literature and future directions. J Dev Behav Pediatr. 2009 Jun;30(3):255-63. doi: 10.1097/DBP.0b013e3181a7ed5a. PMID 19525720
- [Background] Williams DR, Lawrence JA, Davis BA. Racism and Health: Evidence and Needed Research. Annu Rev Public Health. 2019 Apr 1;40:105-125. doi: 10.1146/annurev-publhealth-040218-043750. Epub 2019 Feb 2. PMID 30601726
- [Background] Williams DR, Lawrence JA, Davis BA, Vu C. Understanding how discrimination can affect health. Health Serv Res. 2019 Dec;54 Suppl 2(Suppl 2):1374-1388. doi: 10.1111/1475-6773.13222. Epub 2019 Oct 29. PMID 31663121
- [Background] Coll CG, Magnuson K. Cultural Differences as Sources of Developmental. Handbook of early childhood intervention. 2000;
- [Background] Garcia Coll C, Lamberty G, Jenkins R, McAdoo HP, Crnic K, Wasik BH, Vazquez Garcia H. An integrative model for the study of developmental competencies in minority children. Child Dev. 1996 Oct;67(5):1891-914. PMID 9022222
- [Background] Coll CG, Magnuson K. The psychological experience of immigration: A developmental perspective. Immigration and the family: Research and policy on US immigrants. 1997:91-131.
- [Background] Hepworth AD, Berlin LJ, Martoccio TL, Jones Harden B. Maternal attachment style, sensitivity, and infant obesity risk in low-income, Latino families. Attach Hum Dev. 2021 Feb;23(1):75-89. doi: 10.1080/14616734.2020.1729214. Epub 2020 Mar 4. PMID 32126901
- [Background] Simons SM, Cillessen FH, Hazelzet JA. Determinants of a successful problem list to support the implementation of the problem-oriented medical record according to recent literature. BMC Med Inform Decis Mak. 2016 Aug 2;16:102. doi: 10.1186/s12911-016-0341-0. PMID 27485127
- [Background] McDade TW. Measuring immune function: markers of cell-mediated immunity and inflammation in dried blood spots. In: Ice GH, James GD, eds. Measuring Stress in Humans: A Practical Guide for the Field. Cambridge Univ Press; 2007:181-207. Cambridge Studies in Biological and Evolutionary Anthropology.
- [Background] McDade TW, Williams S, Snodgrass JJ. What a drop can do: dried blood spots as a minimally invasive method for integrating biomarkers into population-based research. Demography. 2007 Nov;44(4):899-925. doi: 10.1353/dem.2007.0038. PMID 18232218
- [Background] Ohri-Vachaspati P, Acciai F, DeLia D, Lloyd K, Yedidia MJ. Accuracy of Parent-Measured and Parent-Estimated Heights and Weights in Determining Child Weight Status. JAMA Pediatr. 2019 Aug 1;173(8):793-795. doi: 10.1001/jamapediatrics.2019.1545. PMID 31206143
- [Background] Woo JG, Daniels SR. Assessment of Body Mass Index in Infancy: It Is Time to Revise Our Guidelines. J Pediatr. 2019 Jan;204:10-11. doi: 10.1016/j.jpeds.2018.09.025. Epub 2018 Oct 5. No abstract available. PMID 30297288
- [Background] Acebo C, Sadeh A, Seifer R, Tzischinsky O, Wolfson AR, Hafer A, Carskadon MA. Estimating sleep patterns with activity monitoring in children and adolescents: how many nights are necessary for reliable measures? Sleep. 1999 Feb 1;22(1):95-103. doi: 10.1093/sleep/22.1.95. PMID 9989370
- [Background] Buckhalt JA, El-Sheikh M, Keller P. Children's sleep and cognitive functioning: race and socioeconomic status as moderators of effects. Child Dev. 2007 Jan-Feb;78(1):213-31. doi: 10.1111/j.1467-8624.2007.00993.x. PMID 17328701
- [Background] Adams EL, Master L, Buxton OM, Savage JS. A longitudinal study of sleep-wake patterns during early infancy using proposed scoring guidelines for actigraphy. Sleep Med. 2019 Nov;63:98-105. doi: 10.1016/j.sleep.2019.05.017. Epub 2019 Jun 8. PMID 31610384
- [Background] Adams EL, Savage JS, Master L, Buxton OM. Time for bed! Earlier sleep onset is associated with longer nighttime sleep duration during infancy. Sleep Med. 2020 Sep;73:238-245. doi: 10.1016/j.sleep.2020.07.003. Epub 2020 Jul 14. PMID 32861189
- [Background] Meltzer LJ, Mindell JA. Impact of a child's chronic illness on maternal sleep and daytime functioning. Arch Intern Med. 2006 Sep 18;166(16):1749-55. doi: 10.1001/archinte.166.16.1749. PMID 16983054
- [Background] Mindell JA, Gould RA, Tikotzky L, Leichman ES, Walters RM. Corrigendum to "Norm-referenced scoring system for the Brief Infant Sleep Questionnaire - Revised (BISQ-R)" [Sleep Med 63 (2019) 106-114]. Sleep Med. 2020 Mar;67:286. doi: 10.1016/j.sleep.2019.12.012. Epub 2020 Feb 6. No abstract available. PMID 32035744
- [Background] Mills-Koonce WR, Cox M. Qualitative ratings for parent-child interaction at 3-48 months of age. (Unpublished coding scales). 2013;
- [Background] Ursache A, Blair C, Granger DA, Stifter C, Voegtline K; Family Life Project Investigators. Behavioral reactivity to emotion challenge is associated with cortisol reactivity and regulation at 7, 15, and 24 months of age. Dev Psychobiol. 2014 Apr;56(3):474-88. doi: 10.1002/dev.21113. Epub 2013 Aug 5. PMID 23918193
- [Background] Leerkes EM, Blankson AN, O'Brien M. Differential effects of maternal sensitivity to infant distress and nondistress on social-emotional functioning. Child Dev. 2009 May-Jun;80(3):762-75. doi: 10.1111/j.1467-8624.2009.01296.x. PMID 19489902
- [Background] Blair C, Ursache A, Mills-Koonce R, Stifter C, Voegtline K, Granger DA; Family Life Project Investigators. Emotional reactivity and parenting sensitivity interact to predict cortisol output in toddlers. Dev Psychol. 2015 Sep;51(9):1271-7. doi: 10.1037/dev0000031. Epub 2015 Jul 20. PMID 26192038
- [Background] Owen M. The NICHD study of early child care mother-infant interaction scales. Unpublished manuscript Dallas, TX: Timberlawn Psychiatric Research Foundation. 1992;
- [Background] NICHD Early Child Care Research Network. Characteristics and quality of child care for toddlers and preschoolers. Applied Developmental Science. 2000;4(3):116-135.
- [Background] Stifter CA, Moding KJ. Understanding and measuring parent use of food to soothe infant and toddler distress: A longitudinal study from 6 to 18 months of age. Appetite. 2015 Dec;95:188-96. doi: 10.1016/j.appet.2015.07.009. Epub 2015 Jul 9. PMID 26164121
- [Background] Goldsmith HH, Rothbart M. The laboratory temperament assessment battery (Locomotor Version 3.1). Madison, WI: University of Wisconsin-Madison. 1999;
- [Background] Carter AS, Briggs-Gowan MJ, Jones SM, Little TD. The Infant-Toddler Social and Emotional Assessment (ITSEA): factor structure, reliability, and validity. J Abnorm Child Psychol. 2003 Oct;31(5):495-514. doi: 10.1023/a:1025449031360. PMID 14561058
- [Background] Carter AS, Briggs-Gowan MJ. ITSEA: Infant-toddler social and emotional assessment examiner's manual. San Antonio, TX: PsychCorp. 2006;